CLINICAL TRIAL: NCT03403374
Title: A Multicenter, Open-label, Single-arm, Study to Evaluate Safety and Tolerability of Repatha in Patients With Homozygous Familial Hypercholesterolemia (HoFH) in India
Brief Title: Safety and Tolerability of Repatha® (Evolocumab) in Indian Participants With Homozygous Familial Hypercholesterolemia
Acronym: RAMAN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20170199; 2020-005111-51 (EudraCT Number)
Record Dates: First submitted 2018-01-03; First posted 2018-01-18 (Actual); Results first posted 2020-11-03 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Homozygous Familial Hypercholesterolemia HoFH
Keywords: Evolocumab; Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — evolocumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evolocumab (Experimental): Evolocumab 420 mg subcutaneous (SC) once monthly (QM) or every 2 weeks (Q2W; for participants on apheresis).
  Interventions: Drug: evolocumab

INTERVENTIONS:
Drug: evolocumab — Administered by SC injection via autoinjector (AI)/pen
  Other Names: Repatha®; EvoMab

SUMMARY:
To describe the safety and tolerability of evolocumab in participants with homozygous familial hypercholesterolemia (HoFH) in India. All participants will receive evolocumab over an 8-week period.

DETAILED DESCRIPTION:
An open-label, multicentre, phase 4 study to describe the safety and tolerability of evolocumab in 30 Indian participants with HoFH. Subjects who meet the inclusion/exclusion criteria and laboratory assessments at screening will be enrolled and will be required to maintain their current lipid-lowering drug therapy throughout the duration of the trial. Participants will receive evolocumab 420 mg subcutaneous (SC) once monthly (QM) and study visits will occur approximately every 4 weeks. Apheresis participants will receive evolocumab 420 mg SC every 2 weeks to correspond with their apheresis schedule. Final administration of evolocumab (for all participants) will occur at week 8. The end of study (EOS) visit will occur at week 12 for all participants.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 12 to ≤ 80 years of age at the time of signing the informed consent
* Diagnosis of HoFH based on low-density lipoprotein cholesterol (LDL-C), familial history and xanthoma
* On a low-fat diet and receiving background lipid-lowering therapy stable for 4 weeks prior to screening and during the time frame of the trial
* Fasting LDL-C at screening > 130 mg/dL (3.4 mmol/L)
* Fasting triglycerides at screening ≤ 400 mg/dL (4.5 mmol/L)

Exclusion Criteria:

* Use of mipomersen or lomitapide within 6 months of screening.
* Known active infection or major hematologic, renal, metabolic, gastrointestinal, hepatic, or endocrine dysfunction
* Currently receiving treatment in another investigational device or drug study, or less than 30 days since ending treatment on another investigational device or drug study(ies)
* Female subject is pregnant or breastfeeding or planning to become pregnant or breastfeed
* Female subjects of childbearing potential unwilling to use an acceptable method of effective contraception
* Subject has known sensitivity to any of the products to be administered during dosing
* History or evidence of any other clinically significant disorder, condition or disease
* Subject has previously received evolocumab or any other proprotein convertase subtilisin/kexin type 9 (PKSK-9)-inhibiting therapy

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-08-04 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2019-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (8):
- India (8):
  - Research Site, Ahmedabad, Gujarat
  - Research Site, Bangalore, Karnataka
  - Research Site, Belagavi, Karnataka
  - Research Site, Kochi, Kerala
  - Research Site, Mumbai, Maharashtra
  - Research Site, Pune, Maharashtra
  - Research Site, New Delhi, National Capital Territory of Delhi
  - Research Site, Lucknow, Uttar Pradesh

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Raal FJ, Hegele RA, Ruzza A, Lopez JAG, Bhatia AK, Wu J, Wang H, Gaudet D, Wiegman A, Wang J, Santos RD. Evolocumab Treatment in Pediatric Patients With Homozygous Familial Hypercholesterolemia: Pooled Data From Three Open-Label Studies. Arterioscler Thromb Vasc Biol. 2024 May;44(5):1156-1164. doi: 10.1161/ATVBAHA.123.320268. Epub 2024 Mar 28. PMID 38545781
- [Derived] Bansal S, Ruzza A, Sawhney J, Kulkarni G, Iyengar S, Mehta V, Hamer A, Wu Y, Raal FJ. Evolocumab in patients with homozygous familial hypercholesterolemia in India. J Clin Lipidol. 2021 Nov-Dec;15(6):814-821. doi: 10.1016/j.jacl.2021.10.003. Epub 2021 Oct 20. PMID 34750081
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 10 study centers in India. The first participant was enrolled on 04 August 2018 and the last participant was enrolled on 29 August 2019.
Period: Overall Study
Arm/Group | Evolocumab
Started | 30
Completed | 29
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Evolocumab
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.2 (13.1)
Age, Customized [Count of Participants; unit: Participants]
  Adolescents (12 - 17 years old) | 13
  Adults (18 - 64 years old) | 16
  Adults (65 - 84 years old) | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 30
Low-Density Lipoprotein Cholesterol (LDL-C) [Mean (Standard Deviation); unit: mg/dL] | 473.5 (135.2)
Apolipoprotein B (ApoB) [Mean (Standard Deviation); unit: mg/dL] | 275.3 (69.1)
Lipoprotein(a) (Lp[a]) [Mean (Standard Deviation); unit: nmol/L] | 201.3 (177.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Includes both serious and non-serious adverse events (AEs). AE: any untoward medical occurrence in a participant. SAE: an AE that meets 1 on the following serious criteria: fatal; life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity; congenital anomaly/birth defect; other medically important serious event. TEAE: any AE starting on or after the first dose of study drug and up to and including 30 days after the end of study drug or the end of study date, whichever is earlier.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Evolocumab
Number analyzed (Participants) | 30
Participants | 10

2. Secondary Outcome: Percent Change From Baseline to Week 12 in Low-Density Lipoprotein Cholesterol (LDL-C)
Time Frame: baseline, week 12
Population: Participants with a baseline and week 12 assessment
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Evolocumab
Number analyzed (Participants) | 29
percent change | -6.4 (22.7)

3. Secondary Outcome: Percent Change From Baseline to Week 12 in Apolipoprotein B (ApoB)
Time Frame: baseline, week 12
Population: Participants with a baseline and week 12 assessment
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Evolocumab
Number analyzed (Participants) | 29
percent change | -6.0 (19.8)

4. Secondary Outcome: Percent Change From Baseline to Week 12 in Lipoprotein(a) (Lp[a])
Time Frame: baseline, week 12
Population: Participants with a baseline and week 12 assessment
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Evolocumab
Number analyzed (Participants) | 29
percent change | -0.2 (26.2)

ADVERSE EVENTS:
Time Frame: All-cause mortality: from enrollment (up to 4 weeks prior to treatment) through end of study (week 12). Serious and other adverse events: from the first dose of study treatment through end of treatment (at week 8) plus 4 weeks (week 12).
Description: All-cause mortality is reported for all participants enrolled in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Arm/Group | Evolocumab
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 2/30
Other Adverse Events (participants affected / at risk) | 8/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Evolocumab (N=30)
Coronary artery disease (Cardiac disorders) | 1
Syncope (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Evolocumab (N=30)
Angina pectoris (Cardiac disorders) | 1
Injection site pain (General disorders) | 1
Injection site swelling (General disorders) | 1
Peripheral swelling (General disorders) | 1
Pyoderma (Infections and infestations) | 1
Varicella (Infections and infestations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Diabetic wound (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2017-08-16): https://cdn.clinicaltrials.gov/large-docs/74/NCT03403374/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-09): https://cdn.clinicaltrials.gov/large-docs/74/NCT03403374/SAP_001.pdf